CLINICAL TRIAL: NCT05943145
Title: Outcomes of Group Dance and Movement Training in Ambulatory MS Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: GroundWorks DanceTheater (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 23-100; 1863441-38-20 (Other Grant/Funding Number: National Endowment for the Arts)
Record Dates: First submitted 2023-05-09; First posted 2023-07-13 (Actual); Last update posted 2023-11-28 (Actual); Status verified 2023-11

CONDITIONS: Multiple Sclerosis
Keywords: dance; movement
MeSH Terms: conditions — Multiple Sclerosis

STUDY DESIGN:
Intervention Model Description: Uncontrolled pre-post intervention study. All participants will complete 14 1-hour dance intervention sessions together as a single group
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Group Dance and Movement Training (Experimental): Group dance and movement sessions
  Interventions: Other: Group Dance and Movement Training

INTERVENTIONS:
Other: Group Dance and Movement Training — Dance movement-based sessions including personalized tasks and imagery, mirroring, and inscription, plus warm-up and cool down practices to ensure physical safety

SUMMARY:
GroundWorks DanceTheater and Cleveland Clinic are partnering to create and offer an initial study of a dance movement-based community program for people with Multiple Sclerosis (MS). The program will address major needs in the MS community including social-emotional well-being, body awareness, and motor function. GroundWorks artists will use a variety of widely accepted movement-based practices with the goal of improving upper and lower body function and overall well-being. By partnering, GroundWorks and Cleveland Clinic hope to encourage more study of the benefits of dance movement-based programming in individuals affected by MS.

DETAILED DESCRIPTION:
GroundWorks DanceTheater and Cleveland Clinic are partnering to design and implement a pilot study of a dance movement-based community program for people with Multiple Sclerosis (MS). The program is aimed at addressing major needs in the MS community including social-emotional well-being, body awareness, and motor function. GroundWorks artists will use a variety of movement-based practices including personalized tasks and imagery, mirroring, and inscription, with the goal of improving upper and lower extremity function, and well-being. Cleveland Clinic will assist GroundWorks in the selection, monitoring, and testing of the participants. Cleveland Clinic will also take the lead with data management and analysis. By partnering, GroundWorks and Cleveland Clinic hope to create a promising program that will lead to further exploring the impact of dance movement-based programming in individuals affected by MS.

ELIGIBILITY:
Inclusion Criteria:

* age 18 to 65 inclusive
* diagnosis of MS (relapsing or progressive form) based on the revised MacDonald Criteria established by a neurologist
* self-reported upper and lower extremity dysfunction
* ability to walk safely without an assistive device (e.g. cane, walker) indoors and outdoors

Exclusion Criteria:

* comorbidity (e.g. cardiac, respiratory, musculoskeletal) representing a contra-indication to the dance movement program
* exacerbation of MS within the past 60 days
* severe cognitive impairment
* clinically significant concern regarding the participant's ability to safely perform study procedures

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2023-04-24 (Actual); Primary Completion 2023-07-14 (Actual); Study Completion 2023-11-27 (Actual)

PRIMARY OUTCOMES:
Timed Up and Go (TUG) | 4 months
  This is a test of functional mobility, commonly used for people with MS. The test measures the time it takes for a person to stand up from a chair, walk 10 feet, turn around, walk back to the chair and sit down.
9 Hole Peg Test (NHPT) | 4 months
  This is a widely used test of upper extremity function in people with MS. The test measures the time it takes for a person to pick up 9 pegs individually and place each one in one of 9 holes on a board and then take each one out, one at a time, and place the pegs back in the container.

SECONDARY OUTCOMES:
Neuro-QOL Positive Affect and Well-Being - Short Form | 4 months
  This is a self-reported quality of life measure which has been validated in people with MS to assess positive affect and well-being.
Neuro-QOL Lower Extremity Function (Mobility) - Short Form | 4 months
  This is a self-reported quality of life measure which has been validated in people with MS to assess mobility.
Neuro-QOL Upper Extremity Function (Fine Motor, ADL) - Short Form | 4 months
  This is a self-reported quality of life measure which has been validated in people with MS to assess fine motor and ADLs.

CONTACTS AND LOCATIONS:
Overall Officials: Francois Bethoux, PhD, Principal Investigator — The Cleveland Clinic
Locations (1):
- Cleveland State University, Cleveland, Ohio, United States

IPD SHARING:
Plan to Share IPD: No